CLINICAL TRIAL: NCT00810199
Title: Randomized Placebo-controlled Study of Two Treatment Strategies Based on Tocilizumab (TCZ) With or Without Methotrexate (MTX) and Possible Addition of Other Disease-modifying Anti-rheumatic Drugs (DMARDs) in Patients...
Brief Title: A Study of Tocilizumab and Methotrexate Treatment Strategies (Adding Tocilizumab to Methotrexate Versus Switching to Tocilizumab) in Patients With Active Rheumatoid Arthritis With Inadequate Response to Prior Methotrexate Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MA21488; 2008-001847-20
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Tocilizumab + Methotrexate (Experimental): Tocilizumab 8 mg/kg (up to 800 mg) intravenous (IV) once every 4 weeks + weekly oral methotrexate continuing at the patient's pre-study dose for 24 weeks. Patients taking oral corticosteroids remained on their pre-study dose (up to 10 mg/day). Week 24 to Week 52 the dose of tocilizumab and methotrexate remained the same. Based on DAS28 assessments, corticosteroid dose was adjusted and disease-modifying antirheumatic drugs (DMARDS) added. Week 52 to Week 104, based on the DAS28 assessment, treatment was adjusted to one of four protocol specified treatment regimens: Treatment tapering, Continued treatment, Treatment intensification or Maintenance treatment. After Week 100, patients who discontinued tocilizumab because of remission were retreated with the last effective dose of tocilizumab or blinded methotrexate if a flare occurred.
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: methotrexate
- Tocilizumab + Placebo (Placebo Comparator): Tocilizumab 8 mg/kg (up to 800 mg) IV once every 4 weeks + weekly oral placebo to methotrexate continuing at the patient's pre-study dose for 24 weeks. Patients taking oral corticosteroids remained on their pre-study dose (up to 10 mg/day). Week 24 to Week 52 the dose of tocilizumab and placebo to methotrexate remained the same. Based on DAS28 assessments, corticosteroid dose was adjusted and disease-modifying antirheumatic drug (DMARDS) added. Week 52 to Week 104, based on the DAS28 assessment, treatment was adjusted to one of four protocol specified treatment regimens: Treatment tapering, Continued treatment, Treatment intensification or Maintenance treatment. After Week 100, patients who discontinued tocilizumab because of remission were retreated with the last effective dose of tocilizumab or blinded placebo to methotrexate if a flare occurred.
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: placebo

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — tocilizumab 8 mg IV every 4 weeks.
  Other Names: RoActemra/Actemra
Drug: methotrexate — Approximately 15-17 mg methotrexate capsule orally once a week.
  Arms: Tocilizumab + Methotrexate
Drug: placebo — Placebo matching methotrexate capsule taken orally once a week.
  Arms: Tocilizumab + Placebo

SUMMARY:
This 2 arm study will compare 2 treatment strategies based on tocilizumab in combination with methotrexate or placebo in patients with moderate to severe rheumatoid arthritis. Patients receiving methotrexate treatment will be randomized to receive either a) tocilizumab 8 mg intravenous (iv) every 4 weeks + methotrexate orally (po) weekly or b) tocilizumab 8 mg iv every 4 weeks + placebo po weekly. After the first 24 weeks of blinded treatment, treatment adjustments (increase or decrease of treatment intensity) may be introduced at intervals, based on response. The anticipated time on study treatment is up to 3 years, and the target sample size is approximately 470 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, ≥ 18 years of age;
* moderate to severe active rheumatoid arthritis (Disease Activity Score (DAS28) > 4.4);
* inadequate response to methotrexate;
* on a stable dose of ≥ 15mg/week methotrexate for at least 6 weeks.

Exclusion Criteria:

* prior treatment with a biologic;
* Rheumatoid arthritis (RA) functional class IV;
* known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections;
* evidence of active malignant disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2009-03; Primary Completion 2010-08 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (120):
- United States (21):
  - Santa Monica, California
  - Upland, California
  - Whittier, California
  - Aventura, Florida
  - Naples, Florida
  - Orange Park, Florida
  - Plantation, Florida
  - Sarasota, Florida
  - South Miami, Florida
  - Tamarac, Florida
  - Eagan, Minnesota
  - Las Vegas, Nevada
  - Mayfield, Ohio
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - West Reading, Pennsylvania
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Spokane, Washington
- Brazil (3):
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - São Paulo, São Paulo
- Croatia (2):
  - Rijeka
  - Zagreb
- Denmark (3):
  - Frederiksberg
  - Hellerup
  - Køge
- Tallinn, Estonia
- France (13):
  - Abbeville
  - Boulogne-Billancourt
  - Brest
  - Échirolles
  - Le Kremlin-Bicêtre
  - Le Mans
  - Marseille
  - Monaco
  - Nantes
  - Nice
  - Paris
  - Pierre-Bénite
  - Vandœuvre-lès-Nancy
- Germany (10):
  - Aachen
  - Berlin
  - Cologne
  - Dresden
  - Erlangen
  - Hamburg
  - Jena
  - München
  - Ratingen
  - Würzburg
- Greece (2):
  - Athens
  - Thessaloniki
- Israel (7):
  - Afula
  - Beersheba
  - Haifa
  - Kfar Saba
  - Ramat Gan
  - Rishon LeZiyyon
  - Tel Aviv
- Italy (5):
  - Ancona
  - Bari
  - Perugia
  - Prato
  - Roma
- Latvia (4):
  - Bauska
  - Daugavpils
  - Liepāja
  - Riga
- Netherlands (5):
  - Amsterdam
  - Leiden
  - Maastricht
  - Nijmegen
  - Utrecht
- Norway (6):
  - Drammen
  - Gjettum
  - Kristiansand
  - Lillehammer
  - Moss
  - Oslo
- Bucharest, Romania
- Russia (14):
  - Barnaul
  - Irkutsk
  - Izhevsk
  - Kazan'
  - Khanty-Mansiysk
  - Kursk
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Tyumen
  - Ufa
  - Ulyanovsk
  - Vladivostok
  - Yekaterinburg
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niška Banja
  - Nova Sad
- Spain (8):
  - Barcelona, Barcelona
  - A Coruña, La Coruña
  - Santiago de Compostela, La Coruña
  - Leganés, Madrid
  - Madrid, Madrid
  - Oviedo, Principality of Asturias
  - Seville, Sevilla
  - Bilbao, Vizcaya
- Sweden (2):
  - Gothenburg
  - Umeå
- Thailand (3):
  - Bangkok
  - Khon Kaen
  - Pathum Thani
- United Kingdom (6):
  - Cannock
  - Glasgow
  - Leeds
  - London
  - Newcastle upon Tyne
  - Norwich

REFERENCES:
- [Result] Dougados M, Kissel K, Sheeran T, Tak PP, Conaghan PG, Mola EM, Schett G, Amital H, Navarro-Sarabia F, Hou A, Bernasconi C, Huizinga TW. Adding tocilizumab or switching to tocilizumab monotherapy in methotrexate inadequate responders: 24-week symptomatic and structural results of a 2-year randomised controlled strategy trial in rheumatoid arthritis (ACT-RAY). Ann Rheum Dis. 2013 Jan;72(1):43-50. doi: 10.1136/annrheumdis-2011-201282. Epub 2012 May 5. PMID 22562983
- [Result] Dougados M, Kissel K, Conaghan PG, Mola EM, Schett G, Gerli R, Hansen MS, Amital H, Xavier RM, Troum O, Bernasconi C, Huizinga TW. Clinical, radiographic and immunogenic effects after 1 year of tocilizumab-based treatment strategies in rheumatoid arthritis: the ACT-RAY study. Ann Rheum Dis. 2014 May;73(5):803-9. doi: 10.1136/annrheumdis-2013-204761. Epub 2014 Jan 28. PMID 24473673
- [Derived] Dougados M, Huizinga TW, Choy EH, Bingham CO 3rd, Aassi M, Bernasconi C. Evaluation of the Disease Activity Score in Twenty-Eight Joints-Based Flare Definitions in Rheumatoid Arthritis: Data From a Three-Year Clinical Trial. Arthritis Care Res (Hoboken). 2015 Dec;67(12):1762-6. doi: 10.1002/acr.22633. PMID 26037777
- [Derived] Huizinga TW, Conaghan PG, Martin-Mola E, Schett G, Amital H, Xavier RM, Troum O, Aassi M, Bernasconi C, Dougados M. Clinical and radiographic outcomes at 2 years and the effect of tocilizumab discontinuation following sustained remission in the second and third year of the ACT-RAY study. Ann Rheum Dis. 2015 Jan;74(1):35-43. doi: 10.1136/annrheumdis-2014-205752. Epub 2014 Aug 28. PMID 25169728

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab + Methotrexate: Tocilizumab 8 mg/kg (up to 800 mg) intravenous (IV) once every 4 weeks + weekly oral methotrexate continuing at the patient's pre-study dose for 24 weeks. Patients taking oral corticosteroids remained on their pre-study dose (up to 10 mg/day). Week 24 to Week 52 the dose of tocilizumab and methotrexate remained the same. Based on DAS28 assessments, corticosteroid dose was adjusted and disease-modifying antirheumatic drug (DMARDS) added. Week 52 to Week 104, based on the DAS28 assessment, treatment was adjusted to one of four protocol specified treatment regimens: Treatment tapering, Continued treatment, Treatment intensification or Maintenance treatment. After Week 100, patients who discontinued tocilizumab because of remission were retreated with the last effective dose of tocilizumab or blinded methotrexate if a flare occurred.
Period: Overall Study
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Started | 279 | 277
Received Study Drug | 277 | 276
Completed Week 24 | 259 | 250
Completed Week 52 | 243 | 229
Completed Week 104 | 222 | 201
Completed | 220 | 195 (Completed=Completed Treatment)
Not Completed | 59 | 82
Not completed — Adverse Event | 24 | 26
Not completed — Death | 4 | 6
Not completed — Withdrew consent | 9 | 12
Not completed — Insufficient therapeutic response | 5 | 14
Not completed — Refused treatment/Did not cooperate | 7 | 7
Not completed — Administrative/Other | 5 | 6
Not completed — Protocol Violation | 2 | 6
Not completed — Failure to return | 1 | 4
Not completed — Did not receive study drug | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline measures are based on the Safety Population and include all randomized participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo | Total
Number analyzed (Participants) | 277 | 276 | 553
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (13.40) | 53.6 (11.91) | 53.3 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 227 | 217 | 444
  Male | 50 | 59 | 109

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Activity Score 28 Joints (DAS28) Remission at Week 24
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. DAS28 Remission is defined as a DAS28 score < 2.6.
Time Frame: Week 24
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Tocilizumab + Methotrexate: Tocilizumab 8 mg/kg intravenous (IV) once every 4 weeks + weekly oral methotrexate continuing at the patient's pre-study dose for 24 weeks.
- Tocilizumab + Placebo: Tocilizumab 8 mg/kg intravenous once every 4 weeks + weekly oral placebo to methotrexate continuing at the patient's pre-study methotrexate dose for 24 weeks.
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Percentage of participants | 40.4 | 34.8
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.2055, Cochran-Mantel-Haenszel — Cochran-Mantel-Haenszel test stratified by region and baseline DAS28 (≤5.5 and >5.5); Odds Ratio (OR) = 1.260, 95% CI 2-sided [0.882 to 1.799]
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.1894, Regression, Logistic — Logistic regression including treatment , region and baseline DAS28; Odds ratio is for Tocilizumab + Methotrexate relative to Tocilizumab + Placebo; Odds Ratio (OR) = 1.270, 95% CI 2-sided [0.889 to 1.814]

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR20) Response
Description: ACR20 response is defined as a ≥ 20% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Baseline, Weeks 24, 52, 104
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Percentage of participants
  Week 24 | 71.5 | 70.3
  Week 52 | 70.8 | 69.2
  Week 104 | 65.7 | 59.4
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.8742, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.6212, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables
Statistical Analysis 3: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 104; Test type: Superiority or Other; p = 0.0963, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables

3. Secondary Outcome: Percentage of Participants With ACR50 Response
Description: ACR50 response is defined as a ≥ 50% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Baseline, Weeks 24, 52, 104
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Percentage of participants
  Week 24 | 45.5 | 40.2
  Week 52 | 50.2 | 55.4
  Week 104 | 52.7 | 46.4
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.2969, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.2215, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables
Statistical Analysis 3: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 104; Test type: Superiority or Other; p = 0.1243, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables

4. Secondary Outcome: Percentage of Participants With ACR70 Response
Description: ACR70 response is defined as a ≥ 70% improvement (reduction) compared with Baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Baseline, Weeks 24, 52, 104
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Percentage of participants
  Week 24 | 24.5 | 25.4
  Week 52 | 31.4 | 31.2
  Week 104 | 34.3 | 29.3
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.6775, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.9976, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables
Statistical Analysis 3: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 104; Test type: Superiority or Other; p = 0.2168, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables

5. Secondary Outcome: Percentage of Participants With ACR90 Response
Description: ACR90 response is defined as a ≥ 90% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: Baseline, Weeks 24, 52, 104
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Percentage of participants
  Week 24 | 5.8 | 5.1
  Week 52 | 12.6 | 11.2
  Week 104 | 11.9 | 9.1
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.8369, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.6528, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables
Statistical Analysis 3: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 104; Test type: Superiority or Other; p = 0.2546, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables

6. Secondary Outcome: Time to First ACR20 Response
Description: Time in days from first administration of study drug until ACR20 response. ACR20 response is defined as a ≥ 20% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: 104 Weeks
Population: Intent-to treat population included all randomized participants who received study drug. Censoring occurred at the last assessment for those completing the study or withdrawing early, if a response was not observed. In calculating ACR response, a last observation carried forward approach is used for missing joint count data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Days | 57.0 [NA to NA] — The minimum and maximum confidence interval was not estimated; insufficient number of participants with events. | 61.0 [57.0 to 84.0]
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.1018, Log Rank

7. Secondary Outcome: Time to First ACR50 Response
Description: Time in days from first administration of study drug until ACR50 response. ACR50 response is defined as a ≥ 50% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate).
Time Frame: 104 Weeks
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Days | 140.0 [113.0 to 142.0] | 143.0 [137.0 to 169.0]
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.7176, Log Rank

8. Secondary Outcome: Time to First ACR70 Response
Description: Time in days from first administration of study drug until ACR70 response. ACR70 response is defined as a ≥ 70% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: 104 Weeks
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Days | 284.0 [225.0 to 327.0] | 307.0 [253.0 to 338.0]
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.8526, Log Rank

9. Secondary Outcome: Time to First ACR90 Response
Description: Time in days from first administration of study drug until ACR90 response. ACR90 response is defined as a ≥ 90% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].
Time Frame: 104 Weeks
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Days | NA [844.0 to NA] — The median was not reached; the rate was < 50%. | NA [986.0 to NA] — The median was not reached; the rate was < 50%.
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.2217, Log Rank

10. Secondary Outcome: Area Under Curve (AUC) DAS28
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. AUC DAS28 was averaged over study days. Analysis of Covariance was adjusted for Baseline DAS28 as a covariate and treatment group and region as fixed factors. Higher calculated AUC values are worse (indicate higher disease activity).
Time Frame: Baseline to Week 24
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug, with data available at Baseline and Week 24.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale*week
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 255 | 246
Score on a scale*week | 3.97 (0.098) | 4.23 (0.092)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.0008, ANCOVA; Baseline DAS28 as a covariate; Mean Difference (Final Values) = -0.26, 95% CI 2-sided [-0.41 to -0.11]

11. Secondary Outcome: Percentage of Participants With Disease Activity Score 28 (DAS28) Remission
Description: as for outcome 1
Time Frame: Week 52
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Tocilizumab + Methotrexate: Tocilizumab 8 mg/kg (up to 800 mg) intravenous (IV) once every 4 weeks + weekly oral methotrexate continuing at the patient's pre-study dose for 24 weeks. Patients taking oral corticosteroids remained on their pre-study dose (up to 10 mg/day). Week 24 to Week 52 the dose of tocilizumab and methotrexate remained the same. Based on DAS28 assessments, corticosteroid dose was adjusted and disease-modifying antirheumatic drug (DMARDS) added.
- Tocilizumab + Placebo: Tocilizumab 8 mg/kg (up to 800 mg) IV once every 4 weeks + weekly oral placebo to methotrexate continuing at the patient's pre-study dose for 24 weeks. Patients taking oral corticosteroids remained on their pre-study dose (up to 10 mg/day). Week 24 to Week 52 the dose of tocilizumab and placebo to methotrexate remained the same. Based on DAS28 assessments, corticosteroid dose was adjusted and disease-modifying antirheumatic drug (DMARDS) added.
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Percentage of participants | 45.5 | 36.6
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.0245, Regression, Logistic; Logistic regression including treatment, region and baseline DAS28; Odds Ratio (OR) = 1.490, 95% CI 2-sided [1.053 to 2.109] — Odds ratio is for Tocilizumab + Methotrexate relative to Tocilizumab + Placebo
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.0258, Cochran-Mantel-Haenszel — Stratified by region and baseline DAS28 (≤ 5.5 and > 5.5); Odds Ratio (OR) = 1.482, 95% CI [1.048 to 2.095]

12. Secondary Outcome: Percentage of Participants With DAS28 Low Disease Activity (LDAS)
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. LDAS is defined as DAS28 ≤ 3.2.
Time Frame: Weeks 24, 52
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Percentage of participants
  Week 24 | 61.7 | 51.4
  Week 52 | 62.5 | 57.2
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.0287, Wald Chi-square; Asymptotic test; parameter estimate is zero
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.2240, Wald Chi-square; Asymptotic test; parameter estimate is zero

13. Secondary Outcome: Change From Baseline in DAS28 Score
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A higher value indicated higher disease activity. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 24, 52
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Score on a scale
  Week 24 | -3.43 (1.326) | -3.21 (1.305)
  Week 52 | -3.74 (1.406) | -3.67 (1.291)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.0497, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.3918, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Percentage of Participants With Good or Moderate European League (EULAR) DAS28 Responses
Description: The DAS28 score is a measure of the patient's disease activity calculated using the tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], patient's global assessment of disease activity [visual analog scale: 0=no disease activity to 100=maximum disease activity] and the erythrocyte sedimentation rate (ESR) for a total possible score of 0 to approximately 10. Scores below 2.6 indicate best disease control and scores above 5.1 indicate worse disease control. A negative change from Baseline indicated improvement.
  European League Against Rheumatism (EULAR) Good response: DAS28 ≤ 3.2 or a change from Baseline < -1.2.
  EULAR Moderate response: DAS28 > 3.2 to ≤ 5.1 or a change from Baseline < -0.6 to ≥ -1.2.
Time Frame: Baseline, 24, 52
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Percentage of participants
  Week 24 | 89.5 | 86.2
  Week 52 | 84.5 | 78.2
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.0019, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.1181, Cochran-Mantel-Haenszel; Region and baseline DAS28 (≤5.5 and >5.5) included as stratification variables

15. Secondary Outcome: Change From Baseline in Swollen Joint Count
Description: 66 joints were assessed for swelling and joints are classified as swollen/not swollen giving a total possible swollen joint count score of 0 to 66. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 24, 52
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Joint count
  Week 24 (n=255,246) | -11.33 (8.042) | -11.74 (9.446)
  Week 52 (n=237,220) | -12.29 (8.796) | -12.25 (8.949)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.7776, Wilcoxon (Mann-Whitney) — P-value is from a 2-sided, Wilcoxon rank-sum test of no difference between the 2 treatment groups in change from baseline
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.8843, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: Change From Baseline in Tender Joint Count
Description: 68 joints are assessed for tenderness and joints are classified as tender/not tender giving a total possible tender joint count score of 0 to 68. A negative change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 24, 52
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Mean (Standard Deviation); unit: Joint count
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Joint count
  Week 24 (n=255,246) | -17.27 (13.358) | -17.00 (13.632)
  Week 52 (n=237,220) | -19.45 (13.471) | -18.97 (12.768)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.9095, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.7179, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity Visual Analog Scale (VAS)
Description: The patients global assessment of disease activity was assessed on a 0 to 100 millimeter (mm) horizontal visual analogue scale (VAS) by the patient. The left-hand extreme of the line equals 0 mm, and was described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 24, 52
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
mm
  Week 24 (n=255,246) | -34.31 (25.677) | -32.42 (24.344)
  Week 52 (n=239,220) | -38.92 (25.590) | -40.94 (26.211)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.3113, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.2931, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity Visual Analog Scale (VAS)
Description: The physician global assessment of disease activity was assessed using a 0 to 100 mm horizontal visual analogue scale (VAS) by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 24, 52
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
mm
  Week 24 (n=249,244) | -40.67 (19.500) | -38.46 (21.654)
  Week 52 (n=232,218) | -44.18 (21.092) | -44.68 (21.400)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.2451, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.8841, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Change From Baseline in Patient Global Assessment of Pain (VAS)
Description: The patient assessed their pain using a 0 to 100 millimeter (mm) horizontal visual analogue scale (VAS). The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". A negative change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 24, 52
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
mm
  Week 24 (n=255,246) | -29.34 (26.639) | -29.75 (24.918)
  Week 52 (239,220) | -33.09 (26.933) | -38.38 (25.537)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.9655, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.0308, Wilcoxon (Mann-Whitney)

20. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR)
Description: Blood was collected for Erythrocyte Sedimentation Rate (ESR) (a test that assesses tissue inflammation) and was analyzed at a local laboratory. ESR was measured in millimeters/hour (mm/hr). A reduction in the level is considered an improvement.
Time Frame: Baseline, Weeks 24, 52
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
mm/hr
  Week 24 (n=255,246) | -30.61 (24.187) | -29.10 (24.518)
  Week 52 (n=238,220) | -31.81 (23.025) | -31.18 (24.527)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.5186, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.7706, Wilcoxon (Mann-Whitney)

21. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP)
Description: Blood was collected for C-Reactive Protein (CRP) (a test for analysis of inflammatory and infectious disorders) and was analyzed at a central laboratory. The serum concentration of CRP was measured in milligrams/deciliter (mg/dL). A reduction in the level is considered an improvement.
Time Frame: Baseline, Weeks 24, 52
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug, with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
mg/dL
  Week 24 (n=252,241) | -1.37 (2.043) | -1.39 (2.206)
  Week 52 (n=236,221) | -1.39 (1.943) | -1.40 (2.216)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.6067, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.6810, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire Disability Index
Description: The Stanford Health Assessment Questionnaire Disability Index (HAQ-DI) is a patient completed questionnaire specific for rheumatoid arthritis, consisting of 20 questions in 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. There are 4 possible responses for each question: 0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do. The score for each of the domains is the highest (worst) score in each domain. A patient must have a domain score for at least 6 of 8 domains to calculate a valid HAQ-DI score which is the sum of domain scores, divided by the number of domains that have a score for a total possible score minimum/maximum 0 (best) to 3 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 24, 52
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug, with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Score on a scale
  Week 24 (n=251,241) | -0.56 (0.666) | -0.55 (0.531)
  Week 52 (n=235,213) | -0.59 (0.713) | -0.67 (0.630)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.9323, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.1448, Wilcoxon (Mann-Whitney)

23. Secondary Outcome: Change From Baseline in Total Genant Modified Sharp Scores (GSS)
Description: Radiographs were taken of each hand and foot at Baseline, Weeks 24, 52 and104 and were evaluated using the Genant modified method according to Sharp. Erosion Score: A total of 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion. Joint Narrowing Score: A total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint). The maximum total erosion score in the hands is 98 and in the feet 42. The maximum scores for joint space narrowing (JSN) in the hands was104 and in the feet 48. The total score was the sum of scores for erosions and JSN. The maximum total modified GSS was 292. A lower number change from Baseline was better. Analysis of covariance model, with Baseline DAS28 as a covariate and treatment and site as fixed factors.
Time Frame: Baseline, Weeks 24, 52, 104
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug, with data available for analysis at Baseline and the given time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Score on a scale
  Week 24 (n= 266,258) | 0.18 (0.161) | 0.35 (0.152)
  Week 52 (n= 269,264) | 0.35 (0.370) | 0.63 (0.350)
  Week 104 (n= 215,202) | 0.35 (0.347) | 0.95 (0.320)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.2034, ANCOVA — Baseline x-ray and DAS28 as covariates and treatment group and region as fixed effects; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.43 to 0.09]
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.3611, ANCOVA — Baseline x-ray and DAS28 as covariates and treatment group and region as fixed effects; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.88 to 0.32]
Statistical Analysis 3: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 104; Test type: Superiority or Other; p = 0.0342, ANCOVA — Baseline x-ray and DAS28 as covariates and treatment group and region as fixed effects; Mean Difference (Final Values) = -0.60, 95% CI 2-sided [-1.16 to -0.05]

24. Secondary Outcome: Change From Baseline in Joint Space Narrowing Score
Description: A total of 13 locations in each hand and wrist and 6 joints in the foot were evaluated for joint narrowing score using a 9-point scale where 0=Normal to 4.0=definite ankylosis (stiffness or fixation of a joint). The maximum scores for joint space narrowing (JSN) in the hands was 104 and in the feet 48 for a total possible score of 0 to 152. A lower change from Baseline indicated a better score. Analysis of covariance model included baseline x-ray and DAS28 as covariates and treatment group and region as fixed effects.
Time Frame: Baseline, Weeks 24, 52, 104
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Score on a scale
  Week 24 (n= 266, 258) | 0.16 (0.121) | 0.19 (0.115)
  Week 52 (n= 269, 264) | 0.45 (0.314) | 0.39 (0.297)
  Week 104 (n= 215, 202) | 0.38 (0.218) | 0.70 (0.201)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.7095, ANCOVA — Baseline x-ray and DAS28 as covariates and treatment group and region as fixed effects; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.23 to 0.16]
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.8147, ANCOVA — Baseline x-ray and DAS28 as covariates and treatment group and region as fixed effects; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.45 to 0.57]
Statistical Analysis 3: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 104; Test type: Superiority or Other; p = 0.0778, ANCOVA — Baseline x-ray and DAS28 as covariates and treatment group and region as fixed effects; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.67 to 0.04]

25. Secondary Outcome: Change From Baseline in Erosion Score
Description: A total of 14 locations in each hand and wrist and 6 joints in the foot were evaluated for erosion using an 8-point scale where 0=Normal to 3.5=very severe erosion. The maximum erosion score in the hands was 98 and in the feet 42 for a total possible score of 0 to 140. A lower number change from Baseline indicated a better score.
Time Frame: Baseline, Weeks 24, 52, 104
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Score on a scale
  Week 24 (n=266,258) | 0.03 (0.077) | 0.15 (0.072)
  Week 52 (n= 269,264) | -0.09 (0.125) | 0.25 (0.118)
  Week 104 (n= 215,202) | -0.03 (0.169) | 0.26 (0.156)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.0441, ANCOVA — Baseline x-ray and DAS28 as covariates and treatment group and region as fixed effects; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.25 to -0.00]
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.0012, ANCOVA — Baseline x-ray and DAS28 as covariates and treatment group and region as fixed effects; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.54 to -0.13]
Statistical Analysis 3: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 104; Test type: Superiority or Other; p = 0.0372, ANCOVA — Baseline x-ray and DAS28 as covariates and treatment group and region as fixed effects; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.56 to -0.02]

26. Secondary Outcome: Percentage of Participants Discontinuing Tocilizumab Due to Remission
Description: The percentage of participants who stopped treatment with tocilizumab due to remission.
Time Frame: Weeks 52, 104
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with non-missing DAS28 assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Percentage of participants
  Week 52 (n=243,231) | 28.4 | 21.6
  Week 104 (n=243,229) | 53.1 | 47.6
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.0694, Cochran-Mantel-Haenszel; Stratified by region and categorical baseline DAS28 (≤ 5.5 and > 5.5); Difference = 6.75, 95% CI 2-sided [-1.02 to 14.52]
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 104; Test type: Superiority or Other; p = 0.1695, Log Rank

27. Secondary Outcome: Percentage of Participants Who Withdrew Due to Lack of Sufficient Therapeutic Response
Description: Lack of Sufficient Therapeutic Response was defined as the patient not responding to the drug as expected.
Time Frame: Up to 3 years
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Percentage of participants | 1.8 | 4.7
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.0496, Cochran-Mantel-Haenszel; Stratified by region and categorical baseline DAS28 (≤ 5.5 and > 5.5); Difference = -2.91, 95% CI [-5.86 to 0.05]

28. Secondary Outcome: Percentage of Participants Who Withdrew Due to Safety Reasons
Description: Safety reasons were defined as adverse events, intercurrent illness or death. An adverse event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. Preexisting conditions that worsened during the study were reported as adverse events.
Time Frame: Up to 3 years
Population: Intent-to-treat population included all randomized participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Percentage of participants | 9.7 | 11.2
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.5188, Cochran-Mantel-Haenszel; Stratified by region and categorical baseline DAS28 (≤ 5.5 and > 5.5); Difference = -1.48, 95% CI 2-sided [-6.59 to 3.62]

29. Secondary Outcome: Change From Baseline in Rheumatoid Arthritis Quality of Life Questionnaire (RAQoL)
Description: The RAQoL is a disease specific patient-reported outcome measure that determines the effect rheumatoid arthritis has on a patient's quality of life consisting of 30 questions that are answered either yes=1 or no=0 for a total possible score ranging from 0 (best) to 30 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 24, 52, 104
Population: Participants from the intent-to-treat Population, all participants who received study drug, with data available for analysis at the given time-point. The RAQoL score was administered in a subset of sites for which the questionnaire was available in the local language.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Score on a scale
  Week 24 (n=146,135) | -6.07 (8.005) | -5.19 (7.064)
  Week 52 (n=132,111) | -7.28 (8.141) | -6.33 (7.691)
  Week 104 (n=87,74) | -6.89 (8.691) | -5.24 (8.899)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 24; Test type: Superiority or Other; p = 0.2652, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Week 52; Test type: Superiority or Other; p = 0.1970, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.1671, Wilcoxon (Mann-Whitney)

30. Secondary Outcome: Change From Baseline in Academic Medical Center (AMC) Linear Disability Scale (ALDS)
Description: The Academic Medical Center (AMC) Linear Disability Score (ALDS) evaluates the participant's ability to perform activities of daily life consisting of 77 questions answered yes or no . The question difficulty and the patient's ability are arranged on a single hierarchical linear scale. ALDS scores range from 10 to 90 with a higher score representing higher functional status. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Weeks 104
Population: Participants from the Intent-to-treat population, all randomized participants who received study drug, with data available for analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 277 | 276
Score on a scale | 2.42 (7.773) | 0.91 (2.099)

31. Secondary Outcome: Area Under the Curve (AUC) From Baseline to Week 24 for ACR Response
Description: ACR response was defined as an improvement (reduction) compared with baseline for both total joint count-68 joints and swollen joint count-66 joints, and for three of five variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) where 0=no pain to 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where: 0=no disease activity to 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate]. Area under the curve for ACR response to Week 24 was averaged over study days. Analysis of covariance model includes treatment group, region and baseline DAS28 (≤ 5.5 and > 5.5) as fixed factors.
Time Frame: Baseline to Week 24
Population: Participants from the intent-to-treat population, all participants who received study drug, with ACR response available for analysis at the time-point. Participants with early withdrawals are not included.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale*day
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 253 | 246
Score on a scale*day | 18.95 (4.220) | 13.74 (3.979)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.1110, ANCOVA; The analysis of covariance model included treatment group, region and baseline DAS28 (≤ 5.5 and > 5.5) as fixed factors; Adjusted Mean Difference (Wald CI) = 5.22, 95% CI 2-sided [-1.20 to 11.64]

32. Secondary Outcome: Area Under the Curve (AUC) From Baseline to Week 52 for ACR Response
Description: ACR response was defined as an improvement (reduction) compared with baseline for both total joint count-68 joints and swollen joint count-66 joints, and for three of five variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) where 0=no pain to 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where: 0=no disease activity to 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant [either C-reactive protein or Erythrocyte Sedimentation Rate].Area under the curve for ACR response to Week 52 averaged over study days. Analysis of covariance model includes treatment group, region and baseline DAS28 (<=5.5 and >5.5) as fixed factors.
Time Frame: Baseline to Week 52
Population: as for outcome 31
Measure: Least Squares Mean (Standard Error); unit: Score on a scale*day
Groups:
- Tocilizumab + Methotrexate: Tocilizumab 8 mg/kg intravenous (IV) once every 4 weeks + weekly oral methotrexate continuing at the patient's pre-study dose for 24 weeks. Patients taking oral corticosteroids remained on their pre-study dose (up to 10 mg/day). Week 24 to Week 52 the dose of tocilizumab and methotrexate remained the same. Based on DAS28 assessments, corticosteroid dose was adjusted and disease-modifying antirheumatic drug (DMARDS) added.
- Tocilizumab + Placebo: Tocilizumab 8 mg/kg intravenous once every 4 weeks + weekly oral placebo to methotrexate continuing at the patient's pre-study methotrexate dose for 24 weeks. Patients taking oral corticosteroids remained on their pre-study dose (up to 10 mg/day). Week 24 to Week 52 the dose of tocilizumab and placebo to methotrexate remained the same. Based on DAS28 assessments, corticosteroid dose was adjusted and disease-modifying antirheumatic drug (DMARDS) added
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 236 | 220
Score on a scale*day | 30.48 (4.901) | 32.59 (4.611)
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.6027, ANCOVA; The analysis of covariance model included treatment group, region and baseline DAS28 (≤ 5.5 and > 5.5) as fixed factors; Adjusted Mean Difference (Wald CI) = -2.11, 95% CI 2-sided [-10.07 to 5.85]

33. Secondary Outcome: Time to Tocilizumab Remission
Description: The time in days from initial study drug treatment to tocilizumab remission that occurred when the patient discontinued treatment with tocilizumab.
Time Frame: 104 Weeks
Population: Participants from the Intent-to-treat population (all randomized participants who received study drug) with data available for this outcome measure. Participants were censored at the last observed value.
Measure: Median (Full Range); unit: Days
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 243 | 229
Days | 645.0 [360 to 855] | 786.0 [351 to 829]
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.1695, Log Rank

34. Secondary Outcome: Time to Drug-Free Remission
Description: The time in days from initial study drug treatment to drug free remission that occurred when the participant was able to discontinue tocilizumab, methotrexate/placebo and open label disease-modifying antirheumatic drugs (DMARDS).
Time Frame: 104 Weeks
Population: as for outcome 33
Measure: Median (Full Range); unit: Days
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 243 | 229
Days | NA [366 to 1121] — Median was not estimated due to the low number of participants with drug-free remission. | NA [365 to 1151] — Median was not estimated due to the low number of participants with drug-free remission.
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.0096, Log Rank

35. Secondary Outcome: Time to Flare After Tocilizumab Remission
Description: The time in days to a flare (recurrence of disease symptoms) after the patient discontinued treatment with tocilizumab.
Time Frame: 104 Weeks
Population: as for outcome 33
Measure: Median (Full Range); unit: Days
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 129 | 109
Days | 113.0 [25 to 400] | 84.0 [1 to 415]
Statistical Analysis 1: Comparison: Tocilizumab + Methotrexate vs Tocilizumab + Placebo; Test type: Superiority or Other; p = 0.0734, Log Rank

36. Secondary Outcome: Time to Restart of Treatment After Discontinuation/Remission
Description: The time in days from treatment discontinuation or remission to the restart of treatment.
Time Frame: 104 Weeks
Population: Participants from the intent-to-treat population, all participants who received study drug, with data available for analysis. Censoring occurred at the last assessment for those completing the study or withdrawing early, if a response had not been observed.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Number analyzed (Participants) | 129 | 109
Days | 113.0 [87.0 to 150.0] | 81.0 [58.0 to 91.0]

ADVERSE EVENTS:
Arm/Group | Tocilizumab + Methotrexate | Tocilizumab + Placebo
Serious Adverse Events (participants affected / at risk) | 49/277 | 48/276
Other Adverse Events (participants affected / at risk) | 189/277 | 179/276
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab + Methotrexate (N=277) | Tocilizumab + Placebo (N=276)
Bronchopneumonia (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 0 | 3
Erysipelas (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Candida endophthalmitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Disseminated tuberculosis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal candidiasis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infected bunion (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Renal abscess (Infections and infestations) | 1 | 0
Scrotal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Typhoid fever (Infections and infestations) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chest pain (General disorders) | 2 | 0
Death (General disorders) | 0 | 1
Device breakage (General disorders) | 0 | 1
Hyperthermia malignant (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 1
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Transaminases increased (Investigations) | 2 | 2
Anxiety (Psychiatric disorders) | 2 | 1
Stress (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Anaphylactoid reaction (Immune system disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Keratitis (Eye disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Colpocele (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab + Methotrexate (N=277) | Tocilizumab + Placebo (N=276)
Nasopharyngitis (Infections and infestations) | 43 | 40
Transaminases increase (Investigations) | 30 | 15
Alanine aminotransferase increased (Investigations) | 33 | 15
Nausea (Gastrointestinal disorders) | 27 | 9
Hypercholesterolemia (Metabolism and nutrition disorders) | 34 | 33
Upper respiratory tract infection (Infections and infestations) | 31 | 25
Urinary tract infection (Infections and infestations) | 23 | 18
Influenza (Infections and infestations) | 18 | 11
Gastroenteritis (Infections and infestations) | 16 | 7
Bronchitis (Infections and infestations) | 17 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 21
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 14 | 15
Diarrhoea (Gastrointestinal disorders) | 20 | 21
Blood cholesterol increased (Investigations) | 12 | 15
Rash (Skin and subcutaneous tissue disorders) | 15 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 16
Headache (Nervous system disorders) | 18 | 21
Leukopenia (Blood and lymphatic system disorders) | 20 | 13
Neutropenia (Blood and lymphatic system disorders) | 15 | 14
Hypertension (Vascular disorders) | 13 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.